CLINICAL TRIAL: NCT05171439
Title: Single-cell Analysis Reveals Surufatinib Mono-therapeutic Efficacy for Second-line Patients With Advanced Hepatocellular Carcinoma: a Single Arm, Open-label, Single Center, Prospective Study
Brief Title: Surufatinib in Advanced Hepatocellular Carcinoma Based on Single-cell Sequencing of Tumor Samples
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Principal Investigator, Beicheng Sun, Director, Hepatobiliary Surgery, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HMPL-012-SPRING-H104
Record Dates: First submitted 2021-12-07; First posted 2021-12-29 (Actual); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: Hepatocellular Carcinoma
Keywords: Surufatinib; single-cell sequencing
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — surufatinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Surufatinib (Experimental): All subjects will receive study treatment in 28-day cycle, Surufatinib 300mg, orally, QD , the treatment will continue until one of the following conditions occurs: progression of disease, death, intolerable toxicity, or the end of study treatment (as other criteria specified in the protocol are met), whichever occurs first.
  Interventions: Drug: Surufatinib

INTERVENTIONS:
Drug: Surufatinib — Surufatinib 300 mg once a day (QD) will be orally administrated on a 28-day cycle
  Other Names: HMPL-012

SUMMARY:
This is a single-arm, single-center, open-label phase II study designed to assess the efficacy of surufatinib in participants with advanced hepatocellular carcinoma based on single-cell sequencing of tumor samples.

DETAILED DESCRIPTION:
This is a single-arm, single-center, open-label phase II study designed to assess the efficacy of surufatinib in participants with advanced hepatocellular carcinoma based on single-cell sequencing of tumor samples. The primary outcome measure of the study is the regulation of immune microenvironment in hepatocellular carcinoma, included the proportion of tumor cells, vascular endothelial cells, and various immune cell clusters (including monocytes, macrophages, mast cells, T cells, B cells, dendritic cells, and neutrophils) in tumor samples before and after treatment with surufatinib, and the expression of related genes. Secondary Efficacy Endpoints include Progression free survival (PFS) (According to RECIST Version 1.1), Objective Response Rate (ORR), Disease Control Rate (DCR), Safety and tolerance will be evaluated by incidence, severity and outcomes of AEs and categorized by severity in accordance with the NCI CTC AE Version 5.0.

ELIGIBILITY:
Inclusion Criteria:

* Ages: 18-75 Years（concluding 18 and 75 Years）;
* Radiologically, histologically or cytologically confirmed hepatocellular carcinoma (HCC) with punctable lesions;
* Barcelona Clinic Liver Cancer stage Category B or C
* ECOG PS 0-1, there was no deterioration within 7 days;
* Liver function status Child-Pugh Class A or B (score≤7)
* Has life expectancy of greater than 12 months；
* HCC patients who received first-line standard chemotherapy (systemic chemotherapy with single or combination drugs such as oxaliplatin) and/or molecular targeted therapies such as sorafenib that failed or were not tolerated;
* Have measurable lesions (according to RECIST 1.1);
* The main organ functions meet the following criteria: (without blood transfusion or any blood component or cell growth factor within 14 days prior to enrollment): Absolute Neutrophil Count (ANC)≥1.5×109/L Platelet Count of ≥100×109/L； Hemoglobin≥90g/L； Total Bilirubin (TBIL)≤1.5 x ULN； ALB≥29 g/L； ALT、AST and ALP≤5 x ULN； Creatinine（Cr）≤1.5×ULN (or creatinine clearance (CCr)≥ 60mL/min); (Only one of albumin and bilirubin in child-Pugh score can be 2 points)
* Male or females patients with reproductive potential must agree to use an effective contraceptive method, for example, double-barrier device, condom, oral or injected birth control medication or intrauterine device, during the study and within 90 days after study treatment discontinuation. All female patients are considered to be fertile, unless the patient had natural menopause or artificial menopause or sterilization (such as hysterectomy, bilateral oophorectomy or ovarian irradiation).
* Good compliance and follow-up

Exclusion Criteria:

* Hepatobiliary duct cell carcinoma and mixed cell carcinoma and fibrolaminar cell carcinoma；
* Patients who intend to undergo liver transplantation (except those who have previously undergone liver transplantation) ;
* Patients who have previously received surufatinib；
* A history of other malignancies within 5 years prior to inclusion, except for cervical carcinoma in situ, basal or squamous cell skin cancer, localized prostate cancer treated with radical surgery, and ductal carcinoma in situ treated with radical surgery;
* Received investigational treatments in other clinical studies within 4 weeks prior to enrollment;
* Use of approved systematic anti-tumor therapy within 4 weeks prior to the first dose, including chemotherapy, biotherapy, targeted therapy (the washout period of small molecular targeted drugs lasts 2 weeks or 5 half-lives, whichever is shorter), hormone therapy, treatments with traditional Chinese medicine (for patients receiving treatments with traditional Chinese medicine with clear anti-tumor indications, for anti-tumor indications clearly specified in the package insert, one-week washout period prior to the first dose is acceptable), etc;
* Received any surgical or invasive treatment or operation (except intravenous catheterization, abdominal puncture and drainage, etc.) within 4 weeks before enrollment;
* International normalized ratio(INR) >1.5 or activated partial thromboplastin time(APTT) >1.5×ULN;
* Presence of clinically significant electrolyte abnormality judged by the investigator;
* Hypertension that is not controlled by the drug, and is defined as: SBP ≥140 mmHg and/or DBP ≥90 mmHg；
* With any diseases or conditions prior to enrollment that affected drug absorption, or patients could not take drugs orally;
* Drugs containing St John's wort taken within 3 weeks prior to the first study treatment, or other strong inducers with CYP3A4 or strong inhibitors taken within two weeks prior to the first study treatment;
* Have a gastrointestinal disease or condition that investigators suspect may affect drug absorption, including, but not limited to, active gastric and duodenal ulcers, ulcerative colitis and other digestive disease, gastrointestinal tumor with active bleeding, or other gastrointestinal conditions that may cause bleeding or perforation, according to the investigator's judgement；
* Patients with evidence or history of obvious bleeding tendency within 3 months before enrollment (>30 ml within 3 months, appeared hematemesis, black dung, hematochezia ) or Hemoptysis (>5 mL of fresh blood within 4 weeks) or a thromboembolic event (including stroke and/or transient ischemic attacks) within 12 months;
* Have clinically significant cardiovascular disease, including but not limited to, acute myocardial infarction; severe/unstable angina pectoris or coronary artery bypass grafting within 6 months prior to enrollment; congestive heart failure according to the New York Heart Association (NYHA) classification ≥ 2; ventricular arrhythmias which needs drug treatment; or left ventricular ejection fraction (LVEF) <50%;
* Active infection or serious infection that is not controlled by drug (≥CTCAE v5.0 Grade 2）;
* History of clinically significant hepatic disease, including, but not limited to, known hepatitis B virus (HBV) infection with HBV DNA positive (copies ≥1×104/ml); known hepatitis C virus infection with HCV RNA positive (copies ≥1×103/m); or liver cirrhosis;
* Mean corrected QT interval (QTc) ≥ 480 msec;
* Occurrence of central nervous system metastatic or known brain metastatic;
* Adverse events (AEs) due to previous anti-tumor therapy has not recovered to Common Terminology Criteria for Adverse Event (CTCAE) ≤Grade 1. Alopecia, lymphocytopenia, and grade ≤2 neurotoxicity due to oxaliplatin are not included;
* Women who are pregnant or lactating;
* With blood transfusion or any blood component or cell growth factor within 14 days prior to enrollment;
* Brachytherapy (i.e., implantation of radioactive seeds) within 60 days before enrollment;
* Urine routine indicates urinary protein ≥ ++, and the 24-hour urine protein quantification is greater than 1.0 g;
* Have any other disease, metabolic disorder, physical examination anomaly, abnormal laboratory result, or any other conditions which, according to judgement of the investigator, renders the patient inappropriate for using the investigational product or affect interpretation of study results.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-09-01 (Estimated); Study Completion 2023-03-01 (Estimated)

PRIMARY OUTCOMES:
Bioinformatics analysis of single-cell sequencing in hepatocellular carcinoma | approximately 1 years
  Analysis of HCC molecular biology information using single cell sequencing technology.

SECONDARY OUTCOMES:
Progression-free Survival (PFS) | approximately 1 years
  A duration from the date of initial treatment to disease progression or death of any cause.
Objective response rate (ORR) | approximately 1 years
  Rate of patients with complete remission (CR) or partial remission (PR) based on RESIST1.1.
Disease control rate (DCR) | approximately 1 years
  Proportion of patients whose tumor volume control (reduced or enlarged) reaches a predetermined value and can maintain a minimum time limit.
adverse events(AE) | approximately 1 years
  adverse events evaluated by the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v5.0.

CONTACTS AND LOCATIONS:
Locations (1):
- Nanjing Drum tower hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No